CLINICAL TRIAL: NCT00615628
Title: Inheritance of Osteosarcoma & Paget's Disease Through Chromosome 18: Examination of Osteosarcoma Tissue Samples From Two Family Members for Loss of Heterozygosity in the Chromosome 18 Region, Genetically Linked With Paget's Disease of Bone
Brief Title: Inheritance of Osteosarcoma & Paget's Disease Through Chromosome 18:
Status: Terminated | Type: Observational
Why Stopped: low enrollment low enrollment
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Timothy Damron, M.D., Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: Osteosarcoma & Paget's Disease; IRB #4168 (Other: IRB number)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Osteosarcoma; Paget's Disease
Keywords: Inheritance of Osteosarcoma & Paget's Disease through Chromosome 18
MeSH Terms: conditions — Osteosarcoma; Osteitis Deformans

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Once a specimen is obtained DNA will be isolated for paraffin-embedded tissue and peripheral blood. Osteosarcoma samples from paraffin embedded, formalin-fixed post-surgical tissue samples will be obtained for the proband and father. Matched normal spamples will be obtained from these individuals as adjacent normal tissue from the post-surgical specimens
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- family members: family members of the proband and father identified

SUMMARY:
Researchers have previously demonstrated loss of heterozygosity in a region on chromosome 18q, associated with osteogenic sarcomas in bone affected by Paget's disease. The loci used in this study are specifically described by those authors as showing loss of heterozygosity in 6 of 7 affected families.

DETAILED DESCRIPTION:
As above, no additional information

ELIGIBILITY:
Inclusion Criteria:

* This is a familial study therefore the only inclusion/exclusion criteria would be that subjects must be a blood relative and over the age of 18.
* The subjects are proband and father along with unaffected blood relatives. Their peripheral blood will act as a control and provide information to delineate the inheritance from the father, as seen in the son.

Exclusion Criteria:

* Not part of the family

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a familial study therefore the only inclusion/exclusion criteria would be that subjects must be a blood relative and over the age of 18. The subjects are proband and father along with unaffected blood relatives. Their peripheral blood will act as a control and provide information to delineate the inheritance from the father, as seen in the son.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2002-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Loss of heterozygosity | January, 2000 through February 2009
  A loss of heterozygosity of a proposed tumor suppressor gene on chromosome 18

CONTACTS AND LOCATIONS:
Overall Officials: Timothy A Damron, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States